CLINICAL TRIAL: NCT00733863
Title: A 52-week,Multi-center,Randomized,Double-blind,Placebo-controlled,Parallel Group Study in Patients With Mild Alzheimer's Disease to Investigate the Safety and Tolerability of Repeated Subcutaneous Injections of CAD106
Brief Title: Safety and Tolerability of Repeated Subcutaneous Injections of CAD106 in Mild Alzheimer's Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCAD106A2201
Record Dates: First submitted 2008-08-08; First posted 2008-08-13 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2010-05

CONDITIONS: Alzheimer Disease
Keywords: Active immunization; Alzheimer disease; Antibody; Central Nervous System Diseases; Neurodegenerative diseases; Vaccine
MeSH Terms: conditions — Alzheimer Disease; Central Nervous System Diseases; Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: CAD106
- 2 (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo
  Arms: 2
Biological: CAD106
  Arms: 1

SUMMARY:
This study will evaluate the safety and tolerability of repeated subcutaneous injections of CAD106 in patients with mild Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Mild Alzheimer's Disease
* Mini-Mental State Examination (MMSE) 20 to 26 at screening, untreated or on stable dose of cholinesterase inhibitor or memantine over the last 6 weeks

Exclusion Criteria:

* Previously participated in an AD vaccine study and received active treatment
* History or presence of an active autoimmune and/or with an acute or chronic inflammation, and/or clinically relevant atopic condition.
* History or presence of seizures and/or cerebrovascular disease.
* Presence of an other neurodegenerative disease and/or psychiatric disorders (with the exception of successfully treated depression)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-07; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability assessments at multiple timepoints including but not limited to screening, baseline, and through the end of the study to Week 52. | 52 weeks

SECONDARY OUTCOMES:
Immune response, cognitive and functional assessments at multiple timepoints including but not limited to baseline and through the end of the study to Week 52. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Principal Investigator — Novartis
Locations (4):
- Centre Hospitalier Universitaire Pellegrin, Bordeaux, France
- Karolinska Universitetssjukhuset Huddinge, Stockholm, Sweden
- NeuroPsychologieZentrum, Basel, Switzerland
- Moorgreen Hospital, Southampton, United Kingdom

REFERENCES:
- [Derived] Farlow MR, Andreasen N, Riviere ME, Vostiar I, Vitaliti A, Sovago J, Caputo A, Winblad B, Graf A. Long-term treatment with active Abeta immunotherapy with CAD106 in mild Alzheimer's disease. Alzheimers Res Ther. 2015 Apr 27;7(1):23. doi: 10.1186/s13195-015-0108-3. eCollection 2015. PMID 25918556